CLINICAL TRIAL: NCT07261553
Title: Adherence to Home-Based Exercise Programs Among Patients With Musculoskeletal Disorders and Its Influencing Factors
Brief Title: Adherence to Home-Based Exercises in Musculoskeletal Disorders
Status: Recruiting | Type: Observational
Sponsor: Konya Beyhekim Training and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Merve Albayrak, Dr., Konya Beyhekim Training and Research Hospital
Other Study IDs: BeyhekimTRHMA2025
Record Dates: First submitted 2025-11-22; First posted 2025-12-03 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-10

CONDITIONS: Exercise Training; Adherence, Treatment; Musculoskeletal Disease; Rehabilitation Exercise; Adherence, Patient; Home Exercise Program
Keywords: Home Exercise Program; adherence; Rehabilitation Exercise; Musculoskeletal Disease; Adherence, Patient
MeSH Terms: conditions — Treatment Adherence and Compliance; Musculoskeletal Diseases; Patient Compliance

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Degenerative: Patients with chronic degenerative musculoskeletal disorders receiving a home exercise program (subcohort)
  Interventions: Other: Home exercise program
- Orthopedic: Patients receiving a home exercise program as part of post-operative orthopedic rehabilitation (subcohort)
  Interventions: Other: Home exercise program
- Neurological: Patients receiving a home exercise program following a neurological condition as part of rehabilitation (subcohort)
  Interventions: Other: Home exercise program

INTERVENTIONS:
Other: Home exercise program — Patients with chronic degenerative musculoskeletal disorders receiving a home exercise program
  Groups: Degenerative
Other: Home exercise program — Patients receiving a home exercise program as part of post-operative orthopedic rehabilitation
  Groups: Neurological
Other: Home exercise program — Patients receiving a home exercise program following a neurological condition as part of rehabilitation
  Groups: Orthopedic

SUMMARY:
Home exercise program is recommended by physicians to patients and their relatives to do at home and It is a treatment option in which the physician describes how to do it. Home workout program to be completed at home to complement and reinforce their program in the clinic It is a personalized set of therapeutic exercises that are taught. There are factors that can change exercise compliance; There are some reasons why some patients adhere to the prescribed home exercise program and others do not.

Adherence to home exercises is a major issue in rehabilitation and the reasons for this are multifactorial; It includes both psychological and specific conditions factors that vary between each individual and these conditions should be taken into account by clinicians in designing personalized exercise programs.

Home exercise programs constitute a fundamental component of rehabilitation and are widely prescribed by physicians support therapeutic gains beyond the clinical environment. These individualized programs aim to maintain functional improvements, reduce symptoms, and promote self-management among individuals with musculoskeletal disorders. Although adherence to home-based exercises is recognized as a key determinant of rehabilitation outcomes, non-adherence remains a persistent challenge. Despite growing emphasis on the importance of exercise compliance, the existing literature provides relatively limited and insufficient evidence regarding the factors that influence adherence across different musculoskeletal conditions, including degenerative, orthopedic, and neurological disorders.

Addressing this gap, the present prospective longitudinal cohort study aims to evaluate adherence to individualized home-based exercise programs among patients with diverse musculoskeletal conditions and to determine whether adherence behaviors differ across diagnostic groups. In addition, the study seeks to identify demographic, clinical, psychosocial, and functional factors associated with exercise compliance. By integrating structured clinical evaluations with validated outcome measures, this study aims not only to clarify the determinants of exercise adherence but also to contribute to the development of more effective, condition-specific strategies to enhance sustained engagement in home-based rehabilitation.

DETAILED DESCRIPTION:
Home exercise programs are recommended by physicians to patients and when appropriate, their caregivers as interventions to be performed outside the clinical setting. In this treatment approach, the physician provides detailed instructions on how the exercises should be carried out. These programs consist of individualized therapeutic exercises designed to be performed at home, with the aim of complementing and reinforcing the interventions delivered in the clinic. Addressing this gap, the present study aims to evaluate adherence to individualized home-based exercise programs among patients with diverse musculoskeletal conditions and to determine whether adherence behaviors differ across diagnostic groups. In addition, the study seeks to identify demographic, clinical, psychosocial, and functional factors associated with exercise compliance. By integrating structured clinical evaluations with validated outcome measures, this study aims not only to clarify the determinants of exercise adherence but also to contribute to the development of more effective, condition-specific strategies to enhance sustained engagement in home-based rehabilitation.

Meeting the inclusion and exclusion criteria; various musculoskeletal diseases; Patients presenting for degenerative, orthopedic or neurological rehabilitation will be included in the study by obtaining written informed consent after an individualized home exercise program after a detailed clinical examination.

Questions such as age, gender, height, weight, education level, employment status, income level and sociodemographic and clinical characteristics of the participants (diagnosis of the disease, duration, comorbidity/cumulative disease score status, medical treatment status, if any, pain/weakness level, functional status) will be recorded.

All patients will receive an individualized home exercise program based on their clinical condition. Exercises will be determined by the physical therapy and rehabilitation physician, taking into account the minimum clinical needs and individual characteristics of the patient. People receiving active physical therapy; will not be included in the study. In terms of content, general physical therapy will consist of exercises, not specific exercises that are rarely practiced or performed by a health professional. The number of sets of exercises per day, how many times they will be done in each set and how many days a week will be defined and recorded. The exercises will be explained to the patient by the physician and the printed paper describing these exercises will be given to the patient.

Three condition-specific subcohorts will be defined: chronic degenerative, orthopedic (post-operative) and neurological patients. Patients in the degenerative, orthopedic, or neurological rehabilitation groups will be provided with a patient-specific home exercise program, and their adherence and adaptations to the program will be evaluated and compared. Patients will do the home-based exercise program for 6 weeks. Patients will undergo both clinical and outcome-based assessments at baseline and again at the completion of the home exercise program (6 weeks).

Among the result criteria; Primary variables; Beck Depression Index (BDI) for mood, Health Assessment Questionnaire (HAQ) for quality of life, Kinesiophobia assessment; Tampa Kinesiophobia Scale, Visual Analog Scale (VAS 0-10), for Activities of Daily Living; Barthel Activities of Daily Living Index Secondary variables; to assess how an individual's health condition affects their daily life for exercise adherence; The Exercise Adherence Rating Scale/Exercise Attitude Questionnarie. All assessments will be evaluated by a group-blind investigator after 6 weeks with clinical examination and a set of evaluation scales/questionnaires. The patients' clinical status, satisfactions, their adherence to exercise therapy, and the factors influencing this adherence will be evaluated. Patients whose diagnosis was established after a detailed examination and for whom an exercise program was prescribed will be included in the study. The decision will be based solely on the patient's ability to perform the exercises and adherence to the inclusion and exclusion criteria. Other factors that could potentially introduce bias, such as education level or the patient's willingness to exercise, will not be considered in determining treatment, in order to minimize selection bias. Patients will be instructed not to take any analgesics within 24 hours prior to the assessment.

ELIGIBILITY:
Inclusion criteria:

* Be 18 years of age or older
* To have a musculoskeletal disease (degenerative, neurological or orthopedic)
* To be given a home exercise program
* To have cognitive and language functions to communicate, to be a volunteer

Exclusion criteria:

* Those with major psychiatric illness
* Those with cognitive dysfunction
* Those with communication disorders, reluctant/reluctant to participate
* Those with any condition other than a primary degenerative, orthopedic, or neurological disease that could significantly affect exercise adherence, including musculoskeletal or systemic disorders (e.g., severe anemia, heart failure, respiratory failure, uncontrolled diabetes, inflammatory rheumatic disease, recent fractures, or active infections).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: * Be 18 years of age or older
  * To have a musculoskeletal disease (degenerative, neurological or orthopedic)
  * To be given a home exercise program
  * To have cognitive and language functions to communicate, to be a volunteer
Sampling Method: Probability Sample
Enrollment: 252 (Estimated)
Dates: Start 2024-07-18 (Actual); Primary Completion 2026-01-30 (Estimated); Study Completion 2026-02-28 (Estimated)

PRIMARY OUTCOMES:
Exercise Adherence Rating Scale | 6th week
  It was developed to evaluate compliance with home exercise programs. The first part (Group A) contains the participant's general information about the exercise program; the second part (Group B; 0-24 points) examines the frequency and sustainability of exercise behaviors; the third part (Group C; 0-40 points) evaluates cognitive and environmental factors affecting exercise adherence. The total score ranges from 0-64, with higher scores indicating greater compliance. The Turkish adaptation, including validation and reliability analysis, was conducted by Korkmaz E in 2019.

SECONDARY OUTCOMES:
VAS | Baseline and 6th week
  VAS ; patients were asked to mark their pain intensity pain activity and rest: 0 no pain; 10 Unbearable/Max. Pain.
  Ranges for the severity of pain and weakness; <3 mild, 3-6 moderate, >6 severe.
Beck Depression Index | Baseline and 6th week
  BDI consists of 21 items related to depressive symptoms such as pessimism, sense of failure, dissatisfaction, feelings of guilt, restlessness, fatigue, decreased appetite, indecision, sleep disturbance, and social withdrawal. Each item contains four levels (0-3) self-evaluation statements that determine a behavior specific to depression . The total maximum score was 63, and a score above 17 indicates an increased risk of depressive states.
Barthel Index | Baseline ve 6th week
  Barthel Index is a general scale developed for independence in activities of daily living. It consists of 10 questions. In the scoring ranging from 0-100 points, 100; best complete independence, 0; the worst refers to absolute dependence.
Tampa Kinesiophobia Scale | Baseline and 6th week
  Tampa Kinesiophobia Scale ; is a 17-question scale developed to measure the fear of movement/re-injury. The scale includes parameters for injury/re-injury and fear-avoidance in work-related activities. A 4-point Likert scoring (1= Strongly disagree, 4= Completely agree) is used in the scale. A total score is calculated after reversing items 4, 8, 12 and 16. The person gets a total score between 17-68. The higher the score of the person on the scale, indicates that kinesiophobia is also high.
Health assessment questionnaire | Baseline and 6th week
  Health assessment questionnaire (HAQ) is the most widely used disease-related, short, easy-to-apply quality of life scale used in clinical research. The scale consists of a total of 21 questions in 8 sub-headings. Each question has a likert type option ranging from 0-3 points. The total score ranges from 0-63. High scores indicate poor (dependent) health.

CONTACTS AND LOCATIONS:
Overall Officials: Ramazan Yilmaz, Study Chair — Konya Beyhekim Training and Research Hospital
Locations (1):
- University of Health Sciences, Konya Beyhekim Training and Research Hospital, Department of Physical Medicine and Rehabilitation, Konya, Turkey 42060, Konya, Konya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No